CLINICAL TRIAL: NCT02386553
Title: An Open-Label Study to Assess the Efficacy, Safety, Tolerability, and Pharmacokinetics of Multiple Doses of ISIS 396443 Delivered Intrathecally to Subjects With Genetically Diagnosed and Presymptomatic Spinal Muscular Atrophy
Brief Title: A Study of Multiple Doses of Nusinersen (ISIS 396443) Delivered to Infants With Genetically Diagnosed and Presymptomatic Spinal Muscular Atrophy
Acronym: NURTURE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 232SM201; 2014-002098-12 (EudraCT Number)
Expanded Access: NCT02865109 (No longer available)
Record Dates: First submitted 2015-02-27; First posted 2015-03-12 (Estimated); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Spinal Muscular Atrophy
Keywords: NURTURE
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — nusinersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (1):
- Nusinersen (Experimental): Nusinersen administered as an intrathecal injection
  Interventions: Drug: Nusinersen

INTERVENTIONS:
Drug: Nusinersen — Solution for intrathecal injection
  Other Names: ISIS 396443; BIIB058; ISIS SMNRx; Spinraza

SUMMARY:
The primary objective of the study is to examine the efficacy of multiple doses of Nusinersen administered intrathecally in preventing or delaying the need for respiratory intervention or death in infants with genetically diagnosed and presymptomatic spinal muscular atrophy (SMA). Secondary objectives of this study are to examine the effects of Nusinersen in infants with genetically diagnosed and presymptomatic SMA.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≤ 6 weeks at first dose.
* Genetic documentation of 5q SMA homozygous gene deletion or mutation or compound heterozygous mutation.
* Genetic documentation of 2 or 3 copies of survival motor neuron 2 (SMN2).
* Ulnar compound muscle action potential (CMAP) ≥ 1 mV at Baseline.
* Gestational age of 37 to 42 weeks for singleton births; gestational age of 34 to 42 weeks for twins.
* Meet additional study related criteria.

Key Exclusion Criteria:

* Hypoxemia (oxygen saturation <96% awake or asleep without any supplemental oxygen or respiratory support).
* Any clinical signs or symptoms at Screening or immediately prior to the first dosing (Day 1) that are, in the opinion of the Investigator, strongly suggestive of SMA.
* Clinically significant abnormalities in hematology or clinical chemistry parameters.
* Treatment with an investigational drug given for the treatment of SMA biological agent, or device. Any history of gene therapy, prior antisense oligonucleotide (ASO) treatment, or cell transplantation.
* Meet additional study related criteria.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 0 Weeks to 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (21):
- United States (11):
  - David Geffen School of Medicine, Los Angeles, California
  - University of California Davis Health System, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Children's Hospital, Orlando, Orlando, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University, New York, New York
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Research Institute, Seattle, Washington
- Australia (2):
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
- Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg, Germany
- Italy (2):
  - Ospedale Pediatrico Bambino Gesù, Rome, Lazio
  - Fondazione Serena Onlus - Centro Clinico Nemo, Milan
- Hamad General Hospital, Doha, Qatar
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (2):
  - Hacettepe University Medical Faculty, Ankara
  - Yeditepe University Medical School Hospital, Istanbul

REFERENCES:
- [Derived] Crawford TO, Swoboda KJ, De Vivo DC, Bertini E, Hwu WL, Finkel RS, Kirschner J, Kuntz NL, Nazario AN, Parsons JA, Pechmann A, Ryan MM, Butterfield RJ, Topaloglu H, Ben-Omran T, Sansone VA, Jong YJ, Shu F, Zhu C, Raynaud S, Lago TR, Paradis AD, Foster R, Chin R, Berger Z; NURTURE Study Group. Continued benefit of nusinersen initiated in the presymptomatic stage of spinal muscular atrophy: 5-year update of the NURTURE study. Muscle Nerve. 2023 Aug;68(2):157-170. doi: 10.1002/mus.27853. Epub 2023 Jul 6. PMID 37409780
- [Derived] Finkel RS, Chiriboga CA, Vajsar J, Day JW, Montes J, De Vivo DC, Yamashita M, Rigo F, Hung G, Schneider E, Norris DA, Xia S, Bennett CF, Bishop KM. Treatment of infantile-onset spinal muscular atrophy with nusinersen: a phase 2, open-label, dose-escalation study. Lancet. 2016 Dec 17;388(10063):3017-3026. doi: 10.1016/S0140-6736(16)31408-8. Epub 2016 Dec 7. PMID 27939059

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the multiple investigative sites from 18 May 2015 to 17 Dec 2024.
Pre-assignment Details: A total of 25 participants diagnosed with Spinal Muscular Atrophy (SMA) were enrolled in the study.
Groups:
- ISIS 396443 2 SMN2 Copies: Participants with 2 survival motor neuron 2 (SMN2) copies received 12 milligrams (mg) nusinersen, intrathecally (IT) on Days 1, 15, 29, 64, 183, 302, 421, 540, 659, 778, 897, 1016, 1135, 1254, 1373, 1492, 1611, 1730, 1849, 1968, 2087, 2206, 2325, 2444, 2563, 2682, and 2801.
- ISIS 396443 3 SMN2 Copies: Participants with 3 SMN2 copies received 12 mg nusinersen, IT on Days 1, 15, 29, 64, 183, 302, 421, 540, 659, 778, 897, 1016, 1135, 1254, 1373, 1492, 1611, 1730, 1849, 1968, 2087, 2206, 2325, 2444, 2563, 2682, and 2801.
Period: Overall Study
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Started | 15 | 10
Completed | 13 | 9
Not Completed | 2 | 1
Not completed — Reason Not Specified | 1 | 1
Not completed — Withdrawal by parent/Guardian | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) set included all participants who received at least 1 dose of ISIS 396443.
Groups:
- ISIS 396443 2 SMN2 Copies: Participants with 2 SMN2 copies received 12 mg nusinersen, IT on Days 1, 15, 29, 64, 183, 302, 421, 540, 659, 778, 897, 1016, 1135, 1254, 1373, 1492, 1611, 1730, 1849, 1968, 2087, 2206, 2325, 2444, 2563, 2682, and 2801.
- Total: Total of all reporting groups
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies | Total
Number analyzed (Participants) | 15 | 10 | 25
Age, Continuous [Mean (Standard Deviation); unit: days] | 19.5 (9.29) | 22.3 (12.45) | 20.6 (10.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 8 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 3 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1 | 0 | 1
  Race: Asian | 1 | 2 | 3
  Race: White | 8 | 6 | 14
  Race: Other | 2 | 1 | 3
  Race: Not Reported Due to Confidentiality Regulations | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Time to Death or Respiratory Intervention
Description: The time was the age of the participant at the first occurrence of either a respiratory intervention or death. Respiratory intervention was defined as invasive or noninvasive ventilation for ≥6 hours/day continuously for 7 or more days OR tracheostomy.
Time Frame: Screening up to Day 2891
Population: The ITT set included all participants who received at least 1 dose of ISIS 396443. Here, 'overall number of participants analyzed' signifies the number of participants with data available for outcome measure analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 5 | 0
months | NA [19.1 to NA] — Median or upper 95% CI not estimable are due to low number of events (i.e. death or respiratory events described above) within the assessed time frame. |

2. Secondary Outcome: Proportion of Participants Developing Clinically Manifested Spinal Muscular Atrophy (SMA)
Description: A participant was considered having clinically manifested SMA if any of the following occurred:
  * Age-adjusted weight <5th percentile or decrease of ≥2 major weight growth curve percentiles (3rd, 5th, 10th, 25th, or 50th) or a percutaneous gastric tube placement for nutritional support
  * Failure to achieve the ability to sit without support
  * Failure to achieve standing with assistance
  * Failure to achieve hands-and-knees crawling
  * Failure to achieve walking with assistance by 24 months of age
  * Failure to achieve standing alone by 24 months of age
  * Failure to achieve walking alone by 24 months of age
Time Frame: At 13 and 24 months of age
Population: The ITT set included all participants who received at least 1 dose of ISIS 396443.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- ISIS 396443 2 SMN2 Copies: Participants with 2 survival motor neuron 2 (SMN2) copies received 12 milligrams (mg) nusinersen, intrathecally (IT) on Days 1, 15, 29, 64, 183, 302, 421, 540, 659, 778, 897, 1016, 1135, 1254, 1373, 1492, 1611, 1730, 1849, 1968, 2087, 2206, 2325, 2444, 2563, 2682, and 2801. test
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 15 | 10
proportion of participants
  13 months of age | 0.67 [0.39 to 0.87] | 0.20 [0.04 to 0.56]
  24 months of age | 0.47 [0.22 to 0.73] | 0 [0.00 to 0.34]

3. Secondary Outcome: Percentage of Participants Alive
Time Frame: Up to 8 years of age
Population: The ITT set included all participants who received at least 1 dose of ISIS 396443.
Measure: Number; unit: percentage of participants
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 15 | 10
percentage of participants | 100 | 100

4. Secondary Outcome: Percentage of Participants Who Attained Motor Milestones Assessed as Part of the Hammersmith Infant Neurological Examination (HINE)
Description: HINE is evaluated in infants between 2-24 months of age. It's a simple, standardized instrument including 26 items assessing different aspects of neurological examinations, such as cranial nerves, posture, movements, tone, and reflexes. In this study, Module 2 of HINE (HINE-2) was assessed, which evaluates 8 developmental milestones (head control, sitting, voluntary grasp, ability to kick, rolling, crawling, standing, and walking) scored on a 3, 4, or 5-point scale, with 0 indicating inability to perform task and score of 2, 3, or 4 indicating full milestone development. Total score is calculated by summing item scores to give maximum possible score of 26. Higher score indicates good neurological function.
Time Frame: Day 700
Population: The ITT set included all participants who received at least 1 dose of ISIS 396443.
Measure: Number; unit: percentage of participants
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 15 | 10
percentage of participants
  First achievement of sitting milestone - Stable sit or Pivots (Rotates) | 100 | 100
  First achievement of standing with support milestone - Stands with support or Stands unaided | 93 | 100
  First achievement of standing unaided milestone - Stands unaided | 73 | 100
  First achievement of walking cruising milestone - Cruising (walks holding on)/Walking independently | 87 | 100
  First achievement of walking milestone - Walking independently | 67 | 100
  First achievement of head control - All the time maintained upright | 100 | 100
  First achievement of voluntary grasp - Pincer grasp | 100 | 100
  First achievement of ability to kick - Touches toes | 100 | 100
  First achievement of rolling - Prone to supine or Supine to prone | 100 | 100
  First achievement of crawling - Crawling on hands and knees | 73 | 100

5. Secondary Outcome: Percentage of Participants Who Attained Motor Milestones as Assessed by World Health Organization (WHO) Criteria
Description: The WHO motor milestones are a set of six milestones in motor development, all of which would be expected to be attained by 24 months of age in healthy children. The individual milestones are: sitting without support, standing with assistance, hands and knees crawling, walking with assistance, standing alone and walking alone.
Time Frame: Baseline up to Day 2891
Population: The ITT set included all participants who received at least 1 dose of ISIS 396443.
Measure: Number; unit: percentage of participants
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 15 | 10
percentage of participants
  First sitting without support milestone achieved using caregiver or site reported dates | 100 | 100
  First hands-and-knees crawling milestone achieved using caregiver or site reported dates | 93 | 100
  First standing with assistance milestone achieved using caregiver or site reported dates | 100 | 100
  First walking with assistance milestone achieved using caregiver or site reported dates | 93 | 100
  First standing alone milestone achieved using caregiver or site reported dates | 93 | 100
  First walking alone milestone achieved using caregiver or site reported dates | 87 | 100

6. Secondary Outcome: Change From Baseline in the Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP INTEND) Motor Function Scale
Description: The CHOP-INTEND test was designed to evaluate the motor skills of infants with signiﬁcant motor weakness. Participants who were ≥2 years were continued to be assessed until a CHOP INTEND maximum score of 64 was achieved. It included 16 items (capturing neck, trunk, and proximal and distal limb strength), nine of which were scored 0, 1, 2, 3, or 4, ﬁve were scored as 0, 2, or 4, one was scored as 0, 1, 2, or 4, and one as 0, 2, 3, or 4 with higher scores indicating greater muscle strength and function. Total score was calculated as the sum of scores for each item. Total score ranged from 0 (worst possible score) and 64 (best possible score). CHOP-INTEND assessments were discontinued once participants achieved a maximum score of 64, so the number of participants with available data points decreased over time.
Time Frame: Baseline, Day 2891
Population: The ITT set included all participants who received at least 1 dose of ISIS 396443. Here 'number analyzed' signifies the number of participants available for analysis at a specified time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 15 | 10
score on a scale
  Baseline | 47.0 (10.04) | 51.9 (6.10)
  Change at Day 2891: number analyzed (Participants) | 2 | 0
  Change at Day 2891 | 29.0 (11.31) |

7. Secondary Outcome: Change From Baseline in Hammersmith Functional Motor Scale - Expanded (HFMSE)
Description: The HFMSE consists of 33 scored activities used to assess motor function in children with SMA. Participants were asked to do a specific activity (such as rolling) and they were then graded on the quality and execution of that movement on a scale of 0=being unable, 1=performed with some compensation, and 2=unaided. The overall score is the sum of the scores for all activities and ranged from 0 to 66. Higher scores indicate increased motor function. Baseline was defined as the time of first HFMSE score after Day 700.
Time Frame: Baseline, Day 2160
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 15 | 10
score on a scale
  Baseline | 34.5 (12.15) | 46.4 (7.44)
  Change at Day 2160: number analyzed (Participants) | 10 | 6
  Change at Day 2160 | 23.5 (5.34) | 22.5 (5.68)

8. Secondary Outcome: Change From Baseline in Weight for Age
Description: The World Health Organization (WHO) child growth standards for participants aged up to 10 years was used to determine the percentiles. WHO Anthro software was used to calculate the percentiles for the given weights of each child. Negative change from baseline indicates low weight for age percentile.
Time Frame: Baseline, Day 2891
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 15 | 10
percentile
  Baseline | 44.04 (31.197) | 34.76 (16.054)
  Change at Day 2891: number analyzed (Participants) | 13 | 9
  Change at Day 2891 | -1.46 (48.041) | 24.49 (40.263)

9. Secondary Outcome: Change From Baseline in Weight for Length
Description: The WHO child growth standards for participants aged up to 10 years was used to determine the percentiles. WHO Anthro software was used to calculate the percentiles for the given weights of each child.
Time Frame: Baseline, Day 1849
Population: The ITT set included all participants who received at least 1 dose of ISIS 396443. Here, 'overall number of participants analyzed' signifies the number of participants with data available for outcome measure analysis. 'number analyzed' signifies the number of participants available for analysis at a specified time point.
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 10 | 6
percentile
  Baseline | 21.63 (22.806) | 45.26 (28.039)
  Change at Day 1849: number analyzed (Participants) | 1 | 0
  Change at Day 1849 | 38.94 (NA) — Since only one participant was evaluable at Day 1849, the standard deviation (SD) could not be estimated. |

10. Secondary Outcome: Change From Baseline in Head Circumference
Time Frame: Baseline, Day 2891
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 15 | 10
centimeter (cm)
  Baseline | 35.59 (2.285) | 36.11 (2.198)
  Change at Day 2891: number analyzed (Participants) | 0 | 1
  Change at Day 2891 |  | 19.00 (NA) — Since only one participant was evaluable at Day 2891, the SD could not be estimated.

11. Secondary Outcome: Change From Baseline in Chest Circumference
Time Frame: Baseline, Day 2891
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 15 | 10
cm
  Baseline | 34.43 (2.724) | 35.25 (2.551)
  Change at Day 2891: number analyzed (Participants) | 0 | 1
  Change at Day 2891 |  | 28.20 (NA) — Since only one participant was evaluable at Day 2891, the SD could not be estimated.

12. Secondary Outcome: Change From Baseline in Head to Chest Circumference Ratio
Description: Negative change from baseline indicates reduction in head-to-chest circumference ratio.
Time Frame: Baseline, Day 2891
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 15 | 10
ratio
  Baseline | 1.036 (0.0537) | 1.027 (0.0595)
  Change at Day 2891: number analyzed (Participants) | 0 | 1
  Change at Day 2891 |  | -0.186 (NA) — Since only one participant was evaluable at Day 2891, the SD could not be estimated.

13. Secondary Outcome: Change From Baseline in Arm Circumference
Time Frame: Baseline, Day 2891
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 15 | 10
cm
  Baseline | 10.85 (1.251) | 10.77 (1.656)
  Change at Day 2891: number analyzed (Participants) | 0 | 1
  Change at Day 2891 |  | 9.40 (NA) — Since only one participant was evaluable at Day 2891, the SD could not be estimated.

14. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE was any unfavorable and unintended sign (including an abnormal assessment such as an abnormal laboratory value), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE was any untoward medical occurrence that at any dose resulted in death, in the view of the Investigator, placed the participant at immediate risk of death, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, resulted in a birth defect.
Time Frame: From the signing of the informed consent form (ICF) up to the end of the study (up to Day 2891)
Population: The ITT set included all participants who received at least 1 dose of ISIS 396443.
Measure: Count of Participants; unit: Participants
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 15 | 10
Participants
  AEs | 15 | 10
  SAEs | 10 | 4

15. Secondary Outcome: Number of Participants With Shifts From Baseline in Clinical Laboratory Parameters (Hematology Parameters)
Description: Hematology parameters included hemoglobin, hematocrit, erythrocytes, platelets, leukocytes, neutrophils, eosinophils, basophils, lymphocytes, and monocytes count. These parameters were flagged as low, normal, or high relative to parameter's normal range or as unknown if no result was available. Here, shift to low indicated values that were normal, high or unknown at baseline and shifted to low values postbaseline. Shift to high indicates values that were normal, low or unknown at baseline and shifted to high postbaseline values.
Time Frame: Baseline up to Day 2891
Population: The ITT set included all participants who received at least 1 dose of ISIS 396443. Here 'number analyzed' signifies the number of participants available for analysis of the specified hematology parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 15 | 10
Participants
  Hemoglobin Shift to Low: number analyzed (Participants) | 13 | 10
  Hemoglobin Shift to Low | 10 | 5
  Hemoglobin Shift to High: number analyzed (Participants) | 13 | 9
  Hemoglobin Shift to High | 3 | 4
  Hematocrit Shift to Low: number analyzed (Participants) | 11 | 10
  Hematocrit Shift to Low | 7 | 7
  Hematocrit Shift to High: number analyzed (Participants) | 13 | 9
  Hematocrit Shift to High | 4 | 4
  Erythrocytes Shift to Low: number analyzed (Participants) | 14 | 9
  Erythrocytes Shift to Low | 3 | 5
  Erythrocytes Shift to High: number analyzed (Participants) | 13 | 9
  Erythrocytes Shift to High | 9 | 3
  Leukocytes Shift to Low: number analyzed (Participants) | 13 | 10
  Leukocytes Shift to Low | 5 | 6
  Leukocytes Shift to High: number analyzed (Participants) | 15 | 9
  Leukocytes Shift to High | 11 | 4
  Neutrophils/Leukocytes Shift to Low: number analyzed (Participants) | 9 | 4
  Neutrophils/Leukocytes Shift to Low | 4 | 2
  Neutrophils/Leukocytes Shift to High: number analyzed (Participants) | 9 | 4
  Neutrophils/Leukocytes Shift to High | 4 | 0
  Eosinophils/Leukocytes Shift to Low | 0 | 0
  Eosinophils/Leukocytes Shift to High: number analyzed (Participants) | 8 | 9
  Eosinophils/Leukocytes Shift to High | 7 | 8
  Basophils/Leukocytes Shift to Low: number analyzed (Participants) | 14 | 10
  Basophils/Leukocytes Shift to Low | 0 | 0
  Basophils/Leukocytes Shift to High: number analyzed (Participants) | 13 | 10
  Basophils/Leukocytes Shift to High | 10 | 9
  Lymphocytes/Leukocytes Shift to Low | 4 | 1
  Lymphocytes/Leukocytes Shift to High: number analyzed (Participants) | 6 | 4
  Lymphocytes/Leukocytes Shift to High | 6 | 4
  Monocytes/Leukocytes Shift to Low: number analyzed (Participants) | 14 | 10
  Monocytes/Leukocytes Shift to Low | 11 | 7
  Monocytes/Leukocytes Shift to High: number analyzed (Participants) | 12 | 6
  Monocytes/Leukocytes Shift to High | 4 | 1
  Neutrophils Shift to Low: number analyzed (Participants) | 9 | 4
  Neutrophils Shift to Low | 2 | 1
  Neutrophils Shift to High: number analyzed (Participants) | 9 | 4
  Neutrophils Shift to High | 3 | 0
  Neutrophils, Segmented Shift to Low | 6 | 4
  Neutrophils, Segmented Shift to High | 9 | 1
  Eosinophils Shift to Low | 0 | 0
  Eosinophils Shift to High: number analyzed (Participants) | 11 | 8
  Eosinophils Shift to High | 11 | 8
  Basophils Shift to Low: number analyzed (Participants) | 15 | 9
  Basophils Shift to Low | 0 | 0
  Basophils Shift to High: number analyzed (Participants) | 14 | 10
  Basophils Shift to High | 4 | 2
  Lymphocytes Shift to Low | 2 | 1
  Lymphocytes Shift to High: number analyzed (Participants) | 14 | 8
  Lymphocytes Shift to High | 11 | 8
  Monocytes Shift to Low | 14 | 10
  Monocytes Shift to High: number analyzed (Participants) | 14 | 6
  Monocytes Shift to High | 4 | 0
  Platelets Shift to Low | 3 | 5
  Platelets Shift to High: number analyzed (Participants) | 10 | 8
  Platelets Shift to High | 9 | 7

16. Secondary Outcome: Number of Participants With Shifts From Baseline in Clinical Laboratory Parameters (Blood Chemistry Parameters)
Description: Blood chemistry parameters included bilirubin (direct and indirect), alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, gamma-glutamyl transferase, creatinine, sodium, potassium, chloride, protein, albumin, calcium, phosphate, glucose, cystatin C, creatine kinase. These parameters were flagged as low, normal, or high relative to parameter's normal range or as unknown if no result was available. Here, shift to low indicated values that were normal, high or unknown at baseline and shifted to low values postbaseline. Shift to high indicates values that were normal, low or unknown at baseline and shifted to high postbaseline values.
Time Frame: Baseline up to Day 2891
Population: The ITT set included all participants who received at least 1 dose of ISIS 396443. Here 'number analyzed' signifies the number of participants available for analysis of the specified blood chemistry parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 15 | 10
Participants
  Bilirubin Shift to Low: number analyzed (Participants) | 14 | 10
  Bilirubin Shift to Low | 14 | 10
  Bilirubin Shift to High: number analyzed (Participants) | 9 | 6
  Bilirubin Shift to High | 2 | 1
  Indirect Bilirubin Shift to Low | 0 | 0
  Indirect Bilirubin Shift to High: number analyzed (Participants) | 8 | 6
  Indirect Bilirubin Shift to High | 1 | 1
  Direct Bilirubin Shift to Low: number analyzed (Participants) | 14 | 10
  Direct Bilirubin Shift to Low | 14 | 10
  Direct Bilirubin Shift to High: number analyzed (Participants) | 13 | 9
  Direct Bilirubin Shift to High | 0 | 1
  Alkaline Phosphatase Shift to Low | 3 | 0
  Alkaline Phosphatase Shift to High: number analyzed (Participants) | 15 | 9
  Alkaline Phosphatase Shift to High | 2 | 5
  Alanine Aminotransferase Shift to Low | 0 | 0
  Alanine Aminotransferase Shift to High: number analyzed (Participants) | 14 | 7
  Alanine Aminotransferase Shift to High | 7 | 2
  Aspartate Aminotransferase Shift to Low | 0 | 0
  Aspartate Aminotransferase Shift to High: number analyzed (Participants) | 14 | 8
  Aspartate Aminotransferase Shift to High | 6 | 2
  Gamma Glutamyl Transferase Shift to Low | 1 | 0
  Gamma Glutamyl Transferase Shift to High | 1 | 0
  Urea Nitrogen Shift to Low: number analyzed (Participants) | 15 | 8
  Urea Nitrogen Shift to Low | 6 | 0
  Urea Nitrogen Shift to High | 0 | 2
  Creatinine Shift to Low: number analyzed (Participants) | 11 | 7
  Creatinine Shift to Low | 5 | 2
  Creatinine Shift to High | 1 | 4
  Sodium Shift to Low: number analyzed (Participants) | 13 | 10
  Sodium Shift to Low | 2 | 0
  Sodium Shift to High | 0 | 1
  Potassium Shift to Low | 0 | 1
  Potassium Shift to High: number analyzed (Participants) | 13 | 7
  Potassium Shift to High | 8 | 3
  Chloride Shift to Low | 0 | 1
  Chloride Shift to High | 0 | 2
  Protein Shift to Low: number analyzed (Participants) | 11 | 8
  Protein Shift to Low | 2 | 5
  Protein Shift to High | 13 | 6
  Albumin Shift to Low: number analyzed (Participants) | 15 | 9
  Albumin Shift to Low | 0 | 0
  Albumin Shift to High: number analyzed (Participants) | 14 | 9
  Albumin Shift to High | 10 | 8
  Bicarbonate Shift to Low: number analyzed (Participants) | 14 | 10
  Bicarbonate Shift to Low | 8 | 7
  Bicarbonate Shift to High | 1 | 0
  Calcium Shift to Low | 3 | 3
  Calcium Shift to High: number analyzed (Participants) | 10 | 9
  Calcium Shift to High | 6 | 8
  Phosphate Shift to Low | 0 | 0
  Phosphate Shift to High: number analyzed (Participants) | 15 | 9
  Phosphate Shift to High | 9 | 4
  Glucose Shift to Low: number analyzed (Participants) | 14 | 10
  Glucose Shift to Low | 7 | 6
  Glucose Shift to High: number analyzed (Participants) | 12 | 8
  Glucose Shift to High | 11 | 7
  Cystatin C Shift to Low: number analyzed (Participants) | 15 | 9
  Cystatin C Shift to Low | 6 | 4
  Cystatin C Shift to High: number analyzed (Participants) | 15 | 9
  Cystatin C Shift to High | 2 | 0
  Creatine Kinase Shift to Low | 0 | 0
  Creatine Kinase Shift to High: number analyzed (Participants) | 9 | 7
  Creatine Kinase Shift to High | 8 | 6

17. Secondary Outcome: Number of Participants With Shifts From Baseline in Clinical Laboratory Parameters (Urinalysis Parameters)
Description: Urinalysis included assessments of specific gravity, pH, protein, glucose, ketones, bilirubin, occult blood, erythrocytes, leukocytes, epithelial cells, bacteria, casts and crystals. These parameters were flagged as low, normal, or high relative to parameter's normal range or as unknown if no result was available. Here, shift to low indicated values that were normal, high or unknown at baseline and shifted to low values postbaseline. Shift to high indicates values that were normal, low or unknown at baseline and shifted to high postbaseline values.
Time Frame: Baseline up to Day 2891
Population: The ITT set included all participants who received at least 1 dose of ISIS 396443. Here 'number analyzed' signifies the number of participants available for analysis of the specified urinalysis parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 15 | 10
Participants
  Specific Gravity Shift to Low: number analyzed (Participants) | 13 | 8
  Specific Gravity Shift to Low | 3 | 1
  Specific Gravity Shift to High | 6 | 5
  pH Shift to Low: number analyzed (Participants) | 14 | 10
  pH Shift to Low | 0 | 1
  pH Shift to High: number analyzed (Participants) | 15 | 9
  pH Shift to High | 3 | 3
  Protein Shift to High/positive: number analyzed (Participants) | 14 | 9
  Protein Shift to High/positive | 13 | 8
  Glucose Shift to High/positive | 1 | 0
  Ketones Shift to High/positive | 9 | 6
  Bilirubin Shift to High/positive | 0 | 0
  Occult Blood Shift to High/positive: number analyzed (Participants) | 15 | 9
  Occult Blood Shift to High/positive | 4 | 2
  Erythrocytes Shift to High/positive | 7 | 1
  Leukocytes Shift to High/positive: number analyzed (Participants) | 12 | 10
  Leukocytes Shift to High/positive | 5 | 4
  Epithelial Cells Shift to High/positive: number analyzed (Participants) | 8 | 3
  Epithelial Cells Shift to High/positive | 5 | 0
  Bacteria Shift to High/positive: number analyzed (Participants) | 7 | 7
  Bacteria Shift to High/positive | 7 | 6
  Casts Shift to High/positive: number analyzed (Participants) | 3 | 3
  Casts Shift to High/positive | 1 | 2
  Crystals Shift to High/positive: number analyzed (Participants) | 2 | 3
  Crystals Shift to High/positive | 1 | 2

18. Secondary Outcome: Number of Participants With Shifts From Baseline in Coagulation Parameters [Activated Partial Thromboplastin Time (aPTT)]
Description: aPTT was evaluated to assess safety. Shift to high measured change in normal, low and unknown values at baseline to high values postbaseline.
Time Frame: Baseline up to Day 2891
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 9 | 8
Participants | 4 | 2

19. Secondary Outcome: Number of Participants With Shifts From Baseline in Coagulation Parameters [Prothrombin Time (PT)]
Description: PT was evaluated to assess safety. Shift to high measured change in normal, low and unknown values at baseline to high values postbaseline.
Time Frame: Baseline up to Day 2891
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 11 | 8
Participants | 7 | 5

20. Secondary Outcome: Number of Participants With Shifts From Baseline in Coagulation Parameters [International Normalized Ratio (INR)]
Description: INR was evaluated to assess safety. Shift to high measured change in normal, low and unknown values at baseline to high values postbaseline.
Time Frame: Baseline up to Day 2891
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 11 | 7
Participants | 4 | 4

21. Secondary Outcome: Percentage of Participants With Clinically Significant Shifts in Electrocardiograms (ECG) Abnormalities
Description: Clinical significance of abnormalities in ECG was determined based on the investigator's discretion. Shift to abnormal indicated values that were normal or unknown at baseline and shifted to abnormal values post-baseline.
Time Frame: Baseline up to Day 2891
Population: The ITT set included all participants who received at least 1 dose of ISIS 396443. Overall number of participants analyzed signifies the number of participants with post-baseline ECG abnormalities.
Measure: Number; unit: percentage of participants
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 12 | 8
percentage of participants | 0 | 0

22. Secondary Outcome: Change From Baseline in Vital Signs (Temperature)
Description: Negative change from baseline indicates reduction in temperature.
Time Frame: Baseline, Day 2891
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 15 | 10
degree Celsius
  Baseline | 36.7 (0.39) | 36.8 (0.44)
  Change at Day 2891: number analyzed (Participants) | 14 | 9
  Change at Day 2891 | 0.0 (0.54) | -0.1 (0.52)

23. Secondary Outcome: Change From Baseline in Vital Signs (Blood Pressure)
Time Frame: Baseline, Day 2891
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 15 | 10
millimeters of mercury (mmHg)
  Baseline-Systolic Blood Pressure | 83.4 (16.40) | 88.1 (17.84)
  Change at Day 2891-Systolic Blood Pressure: number analyzed (Participants) | 14 | 9
  Change at Day 2891-Systolic Blood Pressure | 22.9 (15.29) | 13.6 (15.24)
  Baseline-Diastolic Blood Pressure | 51.1 (17.46) | 50.8 (12.30)
  Change at Day 2891-Diastolic Blood Pressure: number analyzed (Participants) | 14 | 9
  Change at Day 2891-Diastolic Blood Pressure | 12.8 (17.16) | 11.0 (13.07)

24. Secondary Outcome: Change From Baseline in Vital Signs (Heart Rate)
Description: Negative change from baseline indicates reduction in heart rate.
Time Frame: Baseline, Day 2891
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats per minute (beats/min)
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 15 | 9
beats per minute (beats/min)
  Baseline | 141.5 (14.71) | 154.2 (16.55)
  Change at Day 2891: number analyzed (Participants) | 14 | 8
  Change at Day 2891 | -47.2 (20.86) | -62.4 (25.16)

25. Secondary Outcome: Change From Baseline in Vital Signs (Respiratory Rate)
Description: Negative change from baseline indicates reduction in respiratory rate.
Time Frame: Baseline, Day 2891
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: breaths per minute (breaths/min)
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 15 | 10
breaths per minute (breaths/min)
  Baseline | 42.1 (12.17) | 39.8 (13.87)
  Change at Day 2891: number analyzed (Participants) | 14 | 9
  Change at Day 2891 | -21.0 (12.39) | -20.6 (14.43)

26. Secondary Outcome: Number of Participants With Neurological Examination Abnormalities Reported as AEs
Description: Participants with abnormalities in neurological examinations recorded as AEs were reported.
Time Frame: From the signing of the ICF up to the end of the study (up to Day 2891)
Population: The ITT set included all participants who received at least 1 dose of ISIS 396443.
Measure: Count of Participants; unit: Participants
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 15 | 10
Participants
  Muscle contractions involuntary | 8 | 1
  Dysarthria | 7 | 1
  Tremor | 8 | 0
  Hypotonia | 4 | 0
  Areflexia | 2 | 1
  Facial paresis | 2 | 0
  Hyperreflexia | 1 | 1
  Myoclonus | 2 | 0
  Clonus | 1 | 0
  Extensor plantar response | 1 | 0
  Peripheral sensory neuropathy | 1 | 0
  Unresponsive to stimuli | 1 | 0
  Muscular weakness | 9 | 1
  Torticollis | 1 | 1
  Muscle spasms | 0 | 1
  Muscle twitching | 0 | 1
  Trismus | 1 | 0
  Winged scapula | 1 | 0
  Anisocoria | 0 | 1
  Heterophoria | 1 | 0
  Strabismus | 0 | 1
  Vision blurred | 0 | 1
  Automatism | 1 | 0

27. Secondary Outcome: Cerebrospinal Fluid (CSF) Concentration of Nusinersen
Time Frame: Predose on Days 1, 15, 29, 64, 183, 302, 421, 540, 659, 778, 897, 1016, 1135, 1254, 1373, 1492, 1611, 1730, 1849, 1968, 2087, 2206, 2325, 2444, 2563, 2682, 2801
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 15 | 10
nanograms per milliliter (ng/mL)
  Day 1, Pre-dose: number analyzed (Participants) | 14 | 9
  Day 1, Pre-dose | 0.03 (0.00) | 0.03 (0.00)
  Day 15, Pre-dose: number analyzed (Participants) | 14 | 10
  Day 15, Pre-dose | 7.52 (189.00) | 10.22 (285.47)
  Day 29, Pre-dose: number analyzed (Participants) | 14 | 10
  Day 29, Pre-dose | 23.41 (72.04) | 24.56 (85.78)
  Day 64, Pre-dose: number analyzed (Participants) | 12 | 9
  Day 64, Pre-dose | 14.95 (58.06) | 21.33 (63.00)
  Day 183, Pre-dose: number analyzed (Participants) | 14 | 9
  Day 183, Pre-dose | 11.66 (69.60) | 13.85 (54.32)
  Day 302, Pre-dose | 11.34 (54.67) | 10.06 (27.29)
  Day 421, Pre-dose: number analyzed (Participants) | 13 | 10
  Day 421, Pre-dose | 12.20 (66.72) | 10.53 (67.48)
  Day 540, Pre-dose: number analyzed (Participants) | 15 | 9
  Day 540, Pre-dose | 10.23 (38.84) | 9.42 (51.04)
  Day 659, Pre-dose: number analyzed (Participants) | 14 | 10
  Day 659, Pre-dose | 11.91 (42.32) | 10.30 (38.34)
  Day 778, Pre-dose: number analyzed (Participants) | 14 | 10
  Day 778, Pre-dose | 10.87 (54.28) | 11.77 (61.01)
  Day 897, Pre-dose | 11.03 (43.91) | 10.72 (35.90)
  Day 1016, Pre-dose: number analyzed (Participants) | 15 | 9
  Day 1016, Pre-dose | 12.06 (58.41) | 10.65 (39.34)
  Day 1135, Pre-dose | 10.49 (46.05) | 10.87 (36.62)
  Day 1254, Pre-dose: number analyzed (Participants) | 15 | 9
  Day 1254, Pre-dose | 12.88 (47.06) | 11.29 (33.29)
  Day 1373, Pre-dose: number analyzed (Participants) | 14 | 10
  Day 1373, Pre-dose | 11.94 (61.51) | 10.19 (52.12)
  Day 1492, Pre-dose: number analyzed (Participants) | 14 | 8
  Day 1492, Pre-dose | 15.04 (51.20) | 12.71 (92.23)
  Day 1611, Pre-dose: number analyzed (Participants) | 13 | 8
  Day 1611, Pre-dose | 13.46 (40.19) | 13.90 (36.31)
  Day 1730, Pre-dose: number analyzed (Participants) | 9 | 9
  Day 1730, Pre-dose | 13.63 (57.76) | 15.14 (42.12)
  Day 1849, Pre-dose: number analyzed (Participants) | 11 | 9
  Day 1849, Pre-dose | 15.14 (63.15) | 14.19 (42.87)
  Day 1968, Pre-dose: number analyzed (Participants) | 10 | 8
  Day 1968, Pre-dose | 16.52 (67.05) | 17.46 (48.67)
  Day 2087, Pre-dose: number analyzed (Participants) | 12 | 10
  Day 2087, Pre-dose | 15.57 (47.34) | 17.07 (58.91)
  Day 2206, Pre-dose: number analyzed (Participants) | 13 | 9
  Day 2206, Pre-dose | 16.95 (45.86) | 17.16 (46.34)
  Day 2325, Pre-dose: number analyzed (Participants) | 12 | 8
  Day 2325, Pre-dose | 18.27 (59.23) | 20.02 (37.41)
  Day 2444, Pre-dose: number analyzed (Participants) | 13 | 9
  Day 2444, Pre-dose | 16.92 (49.19) | 17.01 (40.87)
  Day 2563, Pre-dose: number analyzed (Participants) | 12 | 9
  Day 2563, Pre-dose | 16.74 (53.14) | 13.37 (85.72)
  Day 2682, Pre-dose: number analyzed (Participants) | 11 | 9
  Day 2682, Pre-dose | 17.42 (44.34) | 16.05 (41.83)
  Day 2801, Pre-dose: number analyzed (Participants) | 13 | 9
  Day 2801, Pre-dose | 17.44 (45.60) | 17.85 (36.35)

28. Secondary Outcome: Plasma Concentration of Nusinersen
Time Frame: Predose on Days 64, 183, 302, 421, 540, 659, 778, 897, 1016, 1135, 1254, 1373, 1492, 1611, 1730, 1849, 1968, 2087, 2206, 2325, 2444, 2563, 2682, 2801 and 4-hour post-dose on Day 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
Number analyzed (Participants) | 15 | 10
ng/ml
  Day 1, 4 hours post-dose: number analyzed (Participants) | 12 | 9
  Day 1, 4 hours post-dose | 391.66 (113.16) | 406.69 (82.92)
  Day 64, Pre-dose | 1.60 (34.52) | 1.56 (46.54)
  Day 183, Pre-dose: number analyzed (Participants) | 13 | 10
  Day 183, Pre-dose | 0.73 (27.03) | 0.81 (19.82)
  Day 302, Pre-dose: number analyzed (Participants) | 14 | 9
  Day 302, Pre-dose | 0.82 (54.28) | 0.81 (21.12)
  Day 421, Pre-dose | 0.78 (39.94) | 0.82 (29.31)
  Day 540, Pre-dose: number analyzed (Participants) | 15 | 9
  Day 540, Pre-dose | 0.72 (29.72) | 0.72 (19.16)
  Day 659, Pre-dose | 0.74 (26.78) | 0.78 (32.51)
  Day 778, Pre-dose | 0.68 (48.37) | 0.81 (23.52)
  Day 897, Pre-dose | 0.71 (34.77) | 0.63 (40.31)
  Day 1016, Pre-dose | 0.69 (38.47) | 0.74 (21.97)
  Day 1135, Pre-dose: number analyzed (Participants) | 13 | 10
  Day 1135, Pre-dose | 0.67 (33.70) | 0.58 (33.78)
  Day 1254, Pre-dose: number analyzed (Participants) | 15 | 8
  Day 1254, Pre-dose | 0.63 (27.16) | 0.60 (24.10)
  Day 1373, Pre-dose | 0.60 (39.79) | 0.59 (17.98)
  Day 1492, Pre-dose: number analyzed (Participants) | 14 | 7
  Day 1492, Pre-dose | 0.69 (40.55) | 0.68 (43.50)
  Day 1611, Pre-dose: number analyzed (Participants) | 13 | 7
  Day 1611, Pre-dose | 0.62 (38.14) | 0.53 (43.12)
  Day 1730, Pre-dose: number analyzed (Participants) | 8 | 9
  Day 1730, Pre-dose | 0.54 (16.13) | 0.53 (30.84)
  Day 1849, Pre-dose: number analyzed (Participants) | 9 | 9
  Day 1849, Pre-dose | 0.47 (52.05) | 0.49 (36.37)
  Day 1968, Pre-dose: number analyzed (Participants) | 10 | 8
  Day 1968, Pre-dose | 0.53 (25.66) | 0.43 (22.96)
  Day 2087, Pre-dose: number analyzed (Participants) | 14 | 9
  Day 2087, Pre-dose | 0.55 (40.43) | 0.47 (31.50)
  Day 2206, Pre-dose: number analyzed (Participants) | 14 | 9
  Day 2206, Pre-dose | 0.43 (43.01) | 0.40 (32.58)
  Day 2325, Pre-dose: number analyzed (Participants) | 12 | 9
  Day 2325, Pre-dose | 0.46 (56.98) | 0.45 (35.19)
  Day 2444, Pre-dose: number analyzed (Participants) | 13 | 9
  Day 2444, Pre-dose | 0.43 (35.15) | 0.51 (17.26)
  Day 2563, Pre-dose: number analyzed (Participants) | 13 | 9
  Day 2563, Pre-dose | 0.38 (61.73) | 0.42 (31.10)
  Day 2682, Pre-dose: number analyzed (Participants) | 12 | 9
  Day 2682, Pre-dose | 0.36 (55.66) | 0.40 (24.48)
  Day 2801, Pre-dose: number analyzed (Participants) | 13 | 9
  Day 2801, Pre-dose | 0.39 (36.16) | 0.35 (65.12)

ADVERSE EVENTS:
Time Frame: From the signing of the ICF up to the end of the study (up to Day 2891)
Description: The ITT set included all participants who received at least 1 dose of ISIS 396443.
Arm/Group | ISIS 396443 2 SMN2 Copies | ISIS 396443 3 SMN2 Copies
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/10
Serious Adverse Events (participants affected / at risk) | 10/15 | 4/10
Other Adverse Events (participants affected / at risk) | 15/15 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ISIS 396443 2 SMN2 Copies (N=15) | ISIS 396443 3 SMN2 Copies (N=10)
Tachycardia (Cardiac disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Coronavirus infection (Infections and infestations) | 1 | 0
Enterovirus infection (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 0
Pneumonia aspiration (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pneumonia pseudomonal (Infections and infestations) | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 2 | 0
Respiratory syncytial virus infection (Infections and infestations) | 2 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Influenza a virus test positive (Investigations) | 1 | 0
Respirovirus test positive (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Feeding disorder (Metabolism and nutrition disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Hyperreflexia (Nervous system disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Medical device change (Surgical and medical procedures) | 1 | 0
Tonsillectomy (Surgical and medical procedures) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ISIS 396443 2 SMN2 Copies (N=15) | ISIS 396443 3 SMN2 Copies (N=10)
Anaemia (Blood and lymphatic system disorders) | 4 | 3
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 5 | 1
Cryptorchism (Congenital, familial and genetic disorders) | 1 | 0
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1 | 0
Epilepsy congenital (Congenital, familial and genetic disorders) | 0 | 1
Hypermobility syndrome (Congenital, familial and genetic disorders) | 0 | 1
Micrognathia (Congenital, familial and genetic disorders) | 2 | 0
Deafness bilateral (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1
Excessive cerumen production (Ear and labyrinth disorders) | 1 | 1
Hyperacusis (Ear and labyrinth disorders) | 1 | 0
Motion sickness (Ear and labyrinth disorders) | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1
Anisocoria (Eye disorders) | 0 | 1
Astigmatism (Eye disorders) | 1 | 1
Dacryostenosis acquired (Eye disorders) | 1 | 0
Eczema eyelids (Eye disorders) | 1 | 0
Eye discharge (Eye disorders) | 1 | 0
Heterophoria (Eye disorders) | 1 | 0
Hypermetropia (Eye disorders) | 0 | 1
Myopia (Eye disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 3 | 1
Strabismus (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Breath odour (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 7 | 1
Dental caries (Gastrointestinal disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 6
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 5 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2
Infantile colic (Gastrointestinal disorders) | 1 | 0
Lip pain (Gastrointestinal disorders) | 0 | 1
Lip swelling (Gastrointestinal disorders) | 1 | 0
Malocclusion (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Teething (Gastrointestinal disorders) | 1 | 2
Tooth loss (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 10 | 5
Application site erythema (General disorders) | 1 | 0
Catheter site pain (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 2
Gait disturbance (General disorders) | 4 | 2
Influenza like illness (General disorders) | 0 | 1
Infusion site bruising (General disorders) | 1 | 0
Infusion site extravasation (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 1
Medical device site rash (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 14 | 8
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Allergy to arthropod bite (Immune system disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Dust allergy (Immune system disorders) | 0 | 1
Food allergy (Immune system disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 2 | 1
Immunodeficiency (Immune system disorders) | 1 | 0
Multiple allergies (Immune system disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 3 | 4
Atypical pneumonia (Infections and infestations) | 1 | 0
Bacterial labyrinthitis (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 4 | 0
Bronchitis (Infections and infestations) | 5 | 1
Bronchitis viral (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Conjunctivitis (Infections and infestations) | 1 | 1
Covid-19 (Infections and infestations) | 5 | 2
Croup infectious (Infections and infestations) | 3 | 0
Cystitis (Infections and infestations) | 1 | 0
Dysentery (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 4 | 2
Ear infection bacterial (Infections and infestations) | 1 | 0
Ear infection staphylococcal (Infections and infestations) | 1 | 0
Enterovirus infection (Infections and infestations) | 1 | 1
Eye infection (Infections and infestations) | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 2
Gastroenteritis viral (Infections and infestations) | 4 | 4
Gastrointestinal viral infection (Infections and infestations) | 1 | 0
Gingivitis (Infections and infestations) | 1 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 3 | 0
Impetigo (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 6 | 4
Labyrinthitis (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 0 | 1
Lice infestation (Infections and infestations) | 1 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 11 | 7
Oral candidiasis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 0 | 2
Otitis externa (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 6 | 5
Otitis media acute (Infections and infestations) | 3 | 1
Otitis media bacterial (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 2 | 1
Pharyngitis streptococcal (Infections and infestations) | 5 | 1
Pneumonia (Infections and infestations) | 7 | 1
Pneumonia aspiration (Infections and infestations) | 3 | 0
Pneumonia moraxella (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 3 | 1
Respiratory tract infection (Infections and infestations) | 3 | 2
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 2
Rhinitis (Infections and infestations) | 3 | 2
Rhinovirus infection (Infections and infestations) | 2 | 0
Rotavirus infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 4 | 3
Sinusitis bacterial (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Stoma site infection (Infections and infestations) | 1 | 0
Streptococcal infection (Infections and infestations) | 1 | 0
Tinea infection (Infections and infestations) | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 11 | 7
Urinary tract infection (Infections and infestations) | 4 | 3
Urinary tract infection bacterial (Infections and infestations) | 1 | 1
Varicella (Infections and infestations) | 2 | 0
Viral infection (Infections and infestations) | 3 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0
Viral rash (Infections and infestations) | 1 | 0
Viral rhinitis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 6 | 3
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 2
Accident (Injury, poisoning and procedural complications) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 3 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 4 | 2
Fall (Injury, poisoning and procedural complications) | 8 | 6
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Lip injury (Injury, poisoning and procedural complications) | 1 | 2
Musculoskeletal procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Nail injury (Injury, poisoning and procedural complications) | 1 | 0
Nasal injury (Injury, poisoning and procedural complications) | 0 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 2 | 4
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 1
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 3 | 5
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0
Radial head dislocation (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 2 | 2
Stoma site hypergranulation (Injury, poisoning and procedural complications) | 1 | 0
Stoma site pain (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Urethral injury (Injury, poisoning and procedural complications) | 0 | 1
Venomous sting (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Adenovirus test positive (Investigations) | 1 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Audiogram abnormal (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Blood calcium increased (Investigations) | 1 | 0
Blood glucose decreased (Investigations) | 0 | 1
Blood iron decreased (Investigations) | 0 | 1
Body temperature increased (Investigations) | 1 | 0
Bone density decreased (Investigations) | 1 | 0
Breath sounds abnormal (Investigations) | 2 | 0
C-reactive protein increased (Investigations) | 2 | 0
Candida test positive (Investigations) | 1 | 0
Carnitine decreased (Investigations) | 1 | 0
Crystal urine present (Investigations) | 1 | 1
Cystatin c increased (Investigations) | 1 | 0
Enterovirus test positive (Investigations) | 1 | 1
Eosinophil count increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Heart rate increased (Investigations) | 1 | 0
Human rhinovirus test positive (Investigations) | 1 | 3
Lymphocyte count increased (Investigations) | 2 | 0
Nerve conduction studies abnormal (Investigations) | 1 | 1
Neutrophil count increased (Investigations) | 2 | 0
Oxygen saturation decreased (Investigations) | 1 | 0
Platelet count increased (Investigations) | 1 | 1
Protein urine present (Investigations) | 1 | 1
Respirovirus test positive (Investigations) | 1 | 0
Sars-cov-2 test positive (Investigations) | 2 | 1
Serratia test positive (Investigations) | 1 | 0
Streptococcus test positive (Investigations) | 1 | 0
Walking distance test abnormal (Investigations) | 1 | 0
Weight decreased (Investigations) | 2 | 1
Weight increased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 2 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0
Feeding disorder (Metabolism and nutrition disorders) | 1 | 0
Feeding intolerance (Metabolism and nutrition disorders) | 1 | 0
Food intolerance (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 2 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0
Lipid metabolism disorder (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Vitamin d deficiency (Metabolism and nutrition disorders) | 1 | 2
Weight gain poor (Metabolism and nutrition disorders) | 2 | 0
Acquired plagiocephaly (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Barrel chest (Musculoskeletal and connective tissue disorders) | 1 | 0
Clubbing (Musculoskeletal and connective tissue disorders) | 1 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 | 0
Growth failure (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint contracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Ligament laxity (Musculoskeletal and connective tissue disorders) | 0 | 1
Lordosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Toe walking (Musculoskeletal and connective tissue disorders) | 2 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 1 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Winged scapula (Musculoskeletal and connective tissue disorders) | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Areflexia (Nervous system disorders) | 2 | 1
Clonus (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 7 | 1
Extensor plantar response (Nervous system disorders) | 1 | 0
Facial paresis (Nervous system disorders) | 2 | 0
Febrile convulsion (Nervous system disorders) | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Gross motor delay (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 3
Hyperreflexia (Nervous system disorders) | 1 | 1
Hypotonia (Nervous system disorders) | 4 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Motor developmental delay (Nervous system disorders) | 2 | 0
Muscle contractions involuntary (Nervous system disorders) | 8 | 1
Myoclonus (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Pleocytosis (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 1
Speech disorder developmental (Nervous system disorders) | 5 | 0
Tremor (Nervous system disorders) | 8 | 0
Unresponsive to stimuli (Nervous system disorders) | 1 | 0
Umbilical granuloma (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Autism spectrum disorder (Psychiatric disorders) | 2 | 0
Automatism (Psychiatric disorders) | 1 | 0
Disturbance in social behaviour (Psychiatric disorders) | 1 | 0
Procedural anxiety (Psychiatric disorders) | 0 | 1
Bladder hypertrophy (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Leukocyturia (Renal and urinary disorders) | 1 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 2 | 0
Vulvovaginal rash (Reproductive system and breast disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 7
Cyanosis central (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary artery dilatation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory muscle weakness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 3
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 3 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 3 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0
Ichthyosis acquired (Skin and subcutaneous tissue disorders) | 0 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Superficial inflammatory dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 2
Aortic dilatation (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Pallor (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2021-10-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT02386553/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT02386553/SAP_001.pdf